CLINICAL TRIAL: NCT02403414
Title: Assessment of Airway in Patients With Acromegaly Undergoing Surgery: Predicting Successful Tracheal Intubation
Brief Title: Assessment of Airway in Patients With Acromegaly for Predicting Successful Tracheal Intubation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Indu Kapoor, Doctor, All India Institute of Medical Sciences
Other Study IDs: IEC/NP-397/14-11-2014
Record Dates: First submitted 2015-03-23; First posted 2015-03-31 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Optical Fibers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Fiberoptic — In the event of failed intubation under direct laryngoscopy, fiberoptic intubation will be performed.

SUMMARY:
Acromegaly is associated with increased risk of difficult intubation and its management. The overall incidence of difficult intubation in patients suffering from acromegaly is four to five times more than those without acromegaly.The difficult intubation scenario in these patients can be managed by various methods ranging from awake fiberoptic intubation to tracheostomy. Difficult tracheal intubation accounts for 17% of respiratory-related injuries and results in significant morbidity and mortality in general population. In patients with acromegaly, inability to mask ventilate or intubate can lead to 28% of all anesthesia related deaths. Therefore, the need and importance of airway assessment in patients with acromegaly cannot be overemphasized. Various tests of airway assessment have to be used to assess difficult airway and tracheal intubation in acromegalics.

The investigators aim to assess the various tests of airway assessment affecting the outcome of patients with acromegaly undergoing pituitary surgery and identify which was best suited.

DETAILED DESCRIPTION:
All the patients of either gender, diagnosed as a case of acromegaly scheduled for pituitary surgery will be enrolled. This observational study will be conducted over a period of 3 years. A written informed consent will be taken from all the patients. The clinical diagnosis will be made on the basis of growth hormone (GH) levels and magnetic resonance imaging (MRI) findings. All patients will be evaluated preoperatively, a day before surgery by an independent observer. Airway assessment for difficult intubation will be performed using Modified Mallampati classification in sitting and supine position followed by mouth opening, upper lip bite test, measurement of thyromental, thyrohyoid, sternomental and hyomental distance. Next the length of upper incisors, presence of receding mandible and neck movement will be checked. An associated history of OSA will also be taken in to account for assessing the difficult intubation followed by OSA grading in acromegalic patients posted for pituitary surgery. In situation of difficult tracheal intubation the fiberoptic intubation would be the preferred choice, which is a gold standard.

General anesthesia will be induced with fentanyl 2µg/kg, propofol 2 mg/kg and rocuronium 1mg/kg. After 90 seconds of mask ventilation, laryngoscopy will be performed with an appropriate sized Macintosh laryngoscope and thereafter Cormac lehane grading will be noted. External laryngeal manipulation (ELM) if carried out will be noted. A standard anesthesia protocol will be followed. After completion of the surgery, neuromuscular blockade will be reversed with neostigmine 0.05mg/kg and glycopyrrolate 0.01mg/kg intravenously. Once the patient follows the verbal command and respiratory parameters are satisfactory, endotracheal tube will be removed. All patients will be shifted to neurosurgical ICU for observation and supportive management.

ELIGIBILITY:
Inclusion Criteria:

* Acromegalic patients undergoing surgery

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with Acromegaly
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Successful tracheal intubation | 10 minutes

SECONDARY OUTCOMES:
Rate of complications | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Indu Kapoor, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- Indu Kapoor, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No